CLINICAL TRIAL: NCT06250608
Title: Evaluation of Cerebral Oxygen Saturation(rSO2) Measurements Between Frontal Lesion Area and Normal Area of Brain by Pulse Oximetry(NIRSITX) Using Near-infrared Spectroscopy in Acute Ischemic Stroke Patients, Prospective, Multi-center, Non-randomized, Open-label, Exploratory Clinical Trial.
Brief Title: Evaluation of rSO2 Between Frontal Lesion Area and Normal Area of Brain by NIRSITX Using NIRS in Acute Ischemic Stroke Patients.
Acronym: fNIRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OBELAB, Inc. (Industry)
Collaborators: Helptrial Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OBE-KMT22-01
Record Dates: First submitted 2024-01-30; First posted 2024-02-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke Patients
Keywords: Stroke; Ischemic Stroke; Acute Ischemic Stroke; Cerebral Oxygen Saturation(rSO2)
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute ischemic stroke patients (Experimental)
  Interventions: Device: Pulse oximeter, NIRSITX

INTERVENTIONS:
Device: Pulse oximeter, NIRSITX — It is a device that non-invasively continuously monitors blood oxygen saturation (rSO2) in localized areas of the brain. This device is attached to patients with symptoms suspected of stroke or diagnosed with stroke to continuously monitor the level of oxygen supply to the brain.

SUMMARY:
The clinical trial is for acute ischemic stroke patients measuring cerebral oxygen saturation (rSO2) values using pulse oximeter of near-infrared spectroscopy in the frontal lesion area and normal area of brain. The purpose of the clinical trial is to compare differences in cerebral oxygen saturation values, and the efficacy and safety are evaluated through additional exploratory clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 19
* Patients diagnosed with acute ischemic stroke within 7 days of symptom onset
* Patient's condition confirmed to have an acute ischemic stroke and also brain blood vessels condition confirmed through brain imaging such as Brain CT/CTA/CT perfusion and Brain MRI/MRA
* Patients voluntarily agree to participate and scheduled to participate in this clinical trial
* Patients willing to comply with the clinical trial protocol

Exclusion Criteria:

* Patients without brain imaging result
* Patients diagnosed with jaundice (hyperbilirubinemia) with abnormal skin color - Patients who find it difficult to wear medical devices for clinical trial on their foreheads
* Patients who has skull fractures of external shape not maintained normal
* Patients who does not agree to participate in this clinical trial
* Patients who are currently participating in another clinical trial or have participated in another clinical trial within 30 days of the screening date
* Patients who is determined from investigator that participating is inappropriate because it may affect the results of the clinical trial or ethically

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of rSO2 values obtained from NIRSITX, a medical device for clinical trials, between the frontal lobe on the side with brain lesions and the frontal lobe on the contralateral side. | Baseline and follow-up (24 hours later)
  The number of study subjects, mean, standard deviation, median, minimum, and maximum are presented as descriptive statistics for the difference and rate of change in rSO2 values obtained from medical equipment for clinical trials between the frontal lobe on the side with the brain lesion and the frontal lobe on the contralateral side. The statistical significance of the change in rSO2 values between two areas is tested using the t-test or Wilcoxon test.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
Investigators must keep confidential all information related to the clinical trial protocol provided by the sponsor or clinical trial monitor. However, exceptions are made when disclosure is requested by the Institutional Review Board, research subjects, or health authorities pursuant to laws or related regulations.
  Personal information of research subjects who participated in clinical trials will be used for up to 6 months after the end of clinical trials, and the collected information will be appropriately managed in accordance with the Personal Information Protection Act. This personal information is not provided to anyone other than the tester.